CLINICAL TRIAL: NCT06525935
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multi-Center Phase 2 Study to Evaluate the Efficacy, Safety, and Tolerability of Once-Weekly CT-388 Administered for 48 Weeks to Participants With Obesity or Overweight With at Least One Weight-Related Comorbidity
Brief Title: A Study of CT-388 in Participants With Obesity or Overweight With at Least One Weight-Related Comorbidity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carmot Therapeutics, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-388-103; XC45526 (Other: Roche Protocol Number)
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1: Placebo (Placebo Comparator): Placebo administered subcutaneously (SC) once weekly.
  Interventions: Drug: Placebo
- Arm 2: CT-388 Dose Level 1 (Low) (Experimental): CT-388 Dose Level 1 administered SC once weekly.
  Interventions: Drug: CT-388
- Arm 3: CT-388 Dose Level 2 (Experimental): CT-388 Dose Level 2 administered SC once weekly.
  Interventions: Drug: CT-388
- Arm 4: CT-388 Dose Level 3 (Experimental): CT-388 Dose Level 3 administered SC once weekly.
  Interventions: Drug: CT-388
- Arm 5: CT-388 Dose Level 4 (Experimental): CT-388 Dose Level 4 administered SC once weekly.
  Interventions: Drug: CT-388
- Arm 6: CT-388 Dose Level 5 (High) (Experimental): CT-388 Dose Level 5 administered SC once weekly.
  Interventions: Drug: CT-388

INTERVENTIONS:
Drug: Placebo — Placebo will be volume- matched and administered subcutaneously (SC) once weekly.
  Arms: Arm 1: Placebo
Drug: CT-388 — CT-388 will be administered subcutaneously (SC) once weekly at the randomized dosing regimen.
  Other Names: RO7795068; RG6640
  Arms: Arm 2: CT-388 Dose Level 1 (Low); Arm 3: CT-388 Dose Level 2; Arm 4: CT-388 Dose Level 3; Arm 5: CT-388 Dose Level 4; Arm 6: CT-388 Dose Level 5 (High)

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, parallel group dose-finding study to evaluate the efficacy and safety of CT-388 at low, middle, and high doses in participants with obesity or who are overweight with at least one weight-related comorbidity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 75 years of age
* Body mass index (BMI) ≥30.0 kg/m2, OR BMI ≥27.0 and <30.0 kg/m2 and previously diagnosed with at least 1 of the following weight-related comorbidities, such as: prediabetes, hypertension, dyslipidemia, obstructive sleep apnea, or cardiovascular disease
* At least one self-reported unsuccessful effort to lose body weight

Exclusion Criteria:

* Prior history/diagnosis/lab evidence of any type of diabetes mellitus (e.g., Type 1, Type 2, gestational), or a history of ketoacidosis or hyperosmolar state
* Self-reported body weight change of >5 kg within 3 months before randomization
* Any unbalanced/extreme diets within 3 months of the screening visit, or plan to be on such diets during the study
* Current or recent participation in an organized weight reduction program
* Current or recent use of any treatment that promotes weight loss or glucose metabolism
* Current or recent use of treatment that may cause weight gain
* Prior or planned surgical treatment for obesity
* Clinically significant or active gastric emptying abnormality, malabsorption, or chronic use of medications that directly affect GI motility
* History of chronic pancreatitis or acute pancreatitis within 6 months before screening
* Have obesity induced by other endocrinologic disorders (e.g., Cushing syndrome) or diagnosed monogenetic or syndromic forms of obesity
* History of major depressive disorder within 2 years of screening, or any history/diagnosis of other severe psychiatric conditions (Note: Prospective participants with depression or anxiety whose disease state, in the opinion of the Investigator, is considered stable and expected to remain stable throughout the course of the study, may be considered for inclusion)
* Family or personal history of medullary thyroid carcinoma
* Serum calcitonin ≥ 20 ng/L
* Women who are pregnant, breastfeeding, or intend to become pregnant, or are of childbearing potential and not using a highly effective contraceptive method

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Percent Change in Body Weight from Baseline to Week 48 | Baseline to Week 48

SECONDARY OUTCOMES:
Percentage of Participants with Body Weight Reduction ≥5%, ≥10%, ≥15%, ≥20%, and ≥25% from Baseline to Week 48 | Baseline and Week 48
Absolute Change in Body Weight (kg) from Baseline to Week 48 | Baseline to Week 48
Percent Change in Body Weight from Baseline to Week 48 by Obesity Class | Baseline to Week 48
Change in Body Mass Index (BMI) from Baseline to Week 48 | Baseline to Week 48
Change in Waist Circumference from Baseline to Week 48 | Baseline to Week 48
Change in Hip Circumference from Baseline to Week 48 | Baseline to Week 48
Change in Waist-to-Hip Ratio from Baseline to Week 48 | Baseline to Week 48
Change in Waist-to-Height Ratio from Baseline to Week 48 | Baseline to Week 48
Change in Glycated Hemoglobin (HbA1c) from Baseline to Week 48 | Baseline to Week 48
Change in Fasting Plasma Glucose from Baseline to Week 48 | Baseline to Week 48
Change in Fasting Insulin from Baseline to Week 48 | Baseline to Week 48
Change in Fasting C-peptide from Baseline to Week 48 | Baseline to Week 48
Change in Fasting Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) from Baseline to Week 48 | Baseline to Week 48
Change in Quantitative Insulin Sensitivity Check Index (QUICKI) from Baseline to Week 48 | Baseline to Week 48
Percentage of Participants with Shift in Glycemic Status from Baseline to Week 48, Based on Fasting Plasma Glucose and HbA1c | Baseline and Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Carmot Therapeutics, Inc., a Member of the Roche Group
Locations (34):
- United States (34):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Central Alabama Research, Homewood, Alabama
  - The Institute for Liver Health II LLC dba Arizona Clinical Trials; Arizona Liver Health, Mesa, Arizona
  - Amicis Research Center - Anaheim, Anaheim, California
  - Ark Clinical-Fountain Valley, Fountain Valley, California
  - Ark Clinical Research - Long Beach, Long Beach, California
  - Velocity Clinical Research - Los Angeles, Los Angeles, California
  - Infinity Clinical Research, Norco, California
  - Amicis Research Center, Northridge, California
  - Prospective Research Innovations Inc., Rancho Cucamonga, California
  - Orange County Research Center, Tustin, California
  - Amicis Research Center - West Hills, West Hills, California
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Louisville Metabolic and Atherosclerosis Research Center (L-MARC), Louisville, Kentucky
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Mercury Street Medical Group, Butte, Montana
  - Neurobehavioral Research, Inc. (NBR), Cedarhurst, New York
  - Lucas Research, Inc, Morehead City, North Carolina
  - Velocity Clinical Research - Cincinnati, Cincinnati, Ohio
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Tribe Clinical Research, Greenville, South Carolina
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Apex Mobile Clinical Research, Bellaire, Texas
  - Velocity Clinical Research - Dallas, Dallas, Texas
  - FutureSearch Trials of Dallas, LLC, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Elevate Clinical, Seabrook, Texas
  - Impact Research Institute, Waco, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - National Clinical Research - Richmond, Inc, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No